CLINICAL TRIAL: NCT07059377
Title: Semaglutide for Smoking Cessation in Patients With Diabetes: A Pilot Randomized Controlled Trial
Brief Title: Semaglutide for Smoking Cessation in Patients With Diabetes
Acronym: GLP1-SC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM74061
Record Dates: First submitted 2025-04-30; First posted 2025-07-10 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2; Nicotine Addiction; Tobacco Dependence
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Tobacco Use Disorder | interventions — semaglutide; Nicotine Replacement Therapy

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Semaglutide + Combination NRT for up to 6 months
  Interventions: Drug: Semaglutide; Drug: Nicotine replacement
- Control (Active Comparator): Combination NRT for up to 6 months
  Interventions: Drug: Nicotine replacement

INTERVENTIONS:
Drug: Semaglutide — Starting dose will be 0.25mg once a week for 4 weeks, then titrated up to 0.5mg once a week. For those requiring additional blood sugar control, the dose may be titrated up to the maximum dose of 2mg once a week. All participants will use this medication for up to 26 weeks
  Arms: Intervention
Drug: Nicotine replacement — Nicotine patch plus short-acting NRT gum or lozenge

SUMMARY:
To assess the feasibility of conducting a randomized controlled trial (RCT) to determine the effectiveness of semaglutide as an adjunct to combination NRT in supporting smoking cessation for patients with diabetes.

DETAILED DESCRIPTION:
Smoking and diabetes are well-established risk factors for cardiovascular disease (CVD) and leading causes of global morbidity and mortality. Glucagon-like peptide-1 receptor agonists (GLP-1 RA) are primarily known for their role in managing diabetes, where they have demonstrated tremendous benefits in glucose control and weight loss. Approximately 12% of adults in the U.S. have ever taken a GLP-1 RA, with 6% currently using these medications. Beyond their primary focus, emerging evidence shows improved clinical outcomes such as Major Adverse Cardiovascular Events (MACE) and Obstructive Sleep Apnea (OSA). Recent research explores the potential role of GLP-1 RA in nicotine addiction. These medications suppress nicotine-induced dopamine release in the nucleus, which supports the exploration of GLP-1 RA therapies for nicotine dependence. Additionally, GLP-1 RA stimulates insulin secretion and reduces energy intake, addressing the common concern of post-cessation weight gain.

While GLP-1 RA have been extensively studied for their effects on weight management, their impact on smoking cessation has only been investigated in a limited number of trials. High-quality evidence is needed using newer and more commonly used GLP-1 RA to assess their effect on smoking cessation and mitigating post-cessation weight gain. We plan to conduct a definitive RCT but need a pilot study to determine feasibility of recruitment, treatment adherence, attrition, and to provide a preliminary estimate of effect size (for sample size calculation).

Research question - Among individuals living with diabetes who smoke, does the addition of GLP-1 RA to combination NRT result in increased smoking cessation at 6-month follow-up?

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older) with type 2 diabetes
* Currently residing in Ontario
* Smoke at least five cigarettes per day and willing to reduce or quit smoking within the next 6 months
* Stable HbA1c ≥7.0% - 10% with no more than a 1% change over the last 3 to 6 months.
* Have not used GLP-1 receptor agonists in the past six months.
* Able to provide informed consent

Exclusion Criteria:

* Pregnant or breastfeeding individuals
* Contraindication to NRT or GLP-1 RA.
* Current daily use of NRT or a GLP1 RA.
* Use of bupropion, cytisine, and varenicline within the last 7 days.
* Use of a DPP-IV inhibitor within the last 7 days.
* Initiation of a new diabetes medication within the last 3 months.
* As per the product monograph, participants with the following diagnoses or disorders will be excluded;
* Personal or family history of medullary thyroid cancer
* Personal or family history of Multiple Endocrine Neoplasia syndrome type 2
* Diabetic ketoacidosis
* Type I diabetes
* Acute pancreatitis or pancreatic cancer
* Acute, chronic or end-stage renal failure
* Tachyarrhythmias
* Unable to engage in follow-up for any reason (for example an acute mental illness, cognitive impairment, unable to speak English or French).
* Other conditions deemed by the study team to interfere with participation or outcomes in the opinion of the study investigator (for example acutely unwell, life expectancy less than 1 year).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Project success | 12 months
  Feasibility will be assessed to provide insights into the potential for a larger trial. Successful completion of this pilot will indicate that a full-scale study is both viable and likely to yield meaningful results. To measure this, the total number of people enrolled will be compared to the total number of people approached to participate.

SECONDARY OUTCOMES:
Smoking status | 6 months
  Participants will be asked if they have quit smoking cigarettesat the 6-month follow-up. This will demonstrate the effectiveness of the pharmacotherapy and GLP-1 products.
Blood glucose score | 6, and 12 months
  The A1c test result is reported as a percentage. The score represents the portion of hemoglobin proteins that are holding glucose. The higher the percentage, the higher blood sugar level an individual has. The range of scores are <5.7% to >10%. Less than 5.7% means no diabetes,5.7% to 6.4% signals prediabetes.
  6.5% or higher usually indicates Type 2 diabetes. HbA1c will be measured at 6 and 12 months in order to measure glycemic control.
Height | 6, and 12 months
  Height will be measured to look for change over time in both groups. It will be recorded in cm.
Weight | 6, and 12 months
  Height will be measured to look for change over time in both groups. It will be recorded in kgs.
Waist circumference | 6, and 12 months
  Height will be measured to look for change over time in both groups. It will be recorded in cm.

IPD SHARING:
Plan to Share IPD: No